CLINICAL TRIAL: NCT06820372
Title: Improving Medication Safety and Prescribing for Individuals Chronic Kidney Disease (CKD) Through the Implementation and Evaluation of an Electronic Drug Dosing and Decision Support Kidney (eDoseCKD) Tool for Nova Scotia Community Pharmacy.
Brief Title: Improving Medication Safety for Kidney Disease with a Digital Drug Dosing Tool in Nova Scotia Community Pharmacy Practice.
Status: Not yet recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Jo-Anne Wilson, Associate Professor, Pharmacy, Faculty of Health, College of Pharmacy, Dalhousie University; Scientific Affiliate, Nova Scotia Health Research and Innovation, Associate Scientist, MSSU, Nova Scotia Health Authority
Other Study IDs: Nova Scotia Health Authority
Record Dates: First submitted 2025-01-31; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5
Keywords: Chronic Kidney Disease; Community Pharmacy; Medication; Tool; mediation safety; decision support algorithms
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Electronic Drug Dosing and Decision Support Kidney (eDoseCKD) Tool — Thirty evidence, expert informed and validated computerized drug decision support algorithms of high risk medications will be utilized by community pharmacists for individuals with an eGFR < 60 ml/min who are on one of the 30 target algorithms. The will be followed up to 3 months to assess effectivess, safety and whether the dose change was maintained.

SUMMARY:
Chronic kidney disease (CKD) is a common condition. It occurs in approximately 7 out of 100 Canadians and is highest in rural settings. The kidneys are responsible for the removal of many drugs from the body. These drugs may require adjustment to avoid buildup. Individuals with CKD also tend to have multiple chronic conditions, are older, and are on many medications. Considering these factors, the risk for unwanted drug effects or harm are high. A recent medication review of a group of Nova Scotians with CKD referred from primary care to a specialist kidney clinic revealed that nearly 20% of high-risk medications should have been dose-adjusted or avoided. In Nova Scotia, community pharmacists' scope of practice now enables them to modify a prescription or prescribe a medication for a chronic condition except CKD. They are in an ideal position to protect or preserve kidney function through appropriate prescribing. Interviews of Nova Scotia community pharmacists in 2022 identified barriers and facilitators for kidney function assessment, medication dose adjustment and prescribing. Key findings indicated the need to develop a tool which would include agreed upon drug dosing based on kidney function, monitoring, medication specific benefits and harms, appropriate alternatives considering drug coverage and ideal medication prescribing to protect and preserve the kidneys. This study objective is to develop, validate, implement, and evaluate an electronic drug dosing and decision support kidney tool (eDoseCKD) in community pharmacy to improve medication safety and optimize kidney health. This project will consist of three phases. Phase one encompassed developing the tool based on evidence, clinician expertise and information learned from a previous study of pharmacists' interviews. Phase two will entailed tool validation or consensus by community pharmacists. In the present study, phase three, the implementation and evaluation of the tool in community pharmacies in Nova Scotia will be undertaken. We aim to answer, will this tool improve medication safety and prescribing in Nova Scotians with CKD? Participating patients will be surveyed to determine satisfaction with quality of care. Participating pharmacists will be interviewed after 6 months to assess barriers to and faciliators for using the computerized decision support alogirthms in community pharmacy practice.

DETAILED DESCRIPTION:
Exploring an Innovative Solution to Optimize Chronic Kidney Disease Management

Chronic kidney disease (CKD) is categorized by a sustained reduction of estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73m2 . The prevalence of CKD in Canada is approximately 12.5 %, representing nearly 3 million adults . In Canadian primary care practices, the prevalence of CKD is 71.9 per 1000 individuals and is highest in rural settings compared to urban settings . Multiple comorbidities, advanced age, and polypharmacy are common in CKD . Many drugs are primarily eliminated by the kidneys and inappropriate dosing can lead to drug accumulation. Considering these factors, the risk for adverse drug events and further harm to kidney function is high in this population .

CKD patients are often exposed to inappropriately prescribed medications which lead to adverse outcomes . In Canada, adverse drug reactions resulting in emergency room visits or hospitalization carry a significant economic burden to the system and health impacts to the individual. A recent Canadian primary care resource outlined key medications to be dose-adjusted or avoided with CKD. The Nova Scotia Health Renal Program published a support tool for primary care providers which included medications to avoid and common drugs requiring renal dose adjustment in those with CKD. Despite the development of these resources, a recent primary care study involving advanced CKD (eGFR less than 60 ml/min/1.73m2) patients in Nova Scotia, found that nearly 20% of high-risk medications that should be dose-adjusted or avoided were not . A possible drawback of these resources is they lack practical suggestions on specific dosing or how to stop a medication, necessary monitoring, appropriate alternatives considering drug coverage or ideal prescribing to protect or preserve kidney function.

Limited progress has unfortunately been made in the past twelve years since the Canadian pharmacotherapy assessment in chronic renal disease (PAIR) instrument revealed that 21% of drug therapy problems in community pharmacy were related to inappropriate use or use of a contraindicated medication . Further, the Canadian Institute for Health information in 2021-2022 reported potentially inappropriate medication prescribing in seniors with rates that were nearly 15% higher in Nova Scotia compared to Canada . This research aims to address the medication prescribing gap that is acute in Nova Scotia through an innovative solution to optimize the resources and capacity of community pharmacists while ensuring safety and quality of medication prescribing in those with CKD.

Cultivating Excellence on the Frontline: Considering the Role of Primary Care Community Pharmacists

According to a recent national survey, more than one in five Canadians do not have a primary care provider. In Atlantic Canada, the proportion of individuals without a prescriber (31%) was more than double that of Ontario (13%). In February of 2023, approximately 135, 000 Nova Scotians were without a primary care provider. Benefits of community pharmacists as prescribers have been highlighted particularly during the COVID-19 pandemic. Pharmacists' scope of practice in Nova Scotia has expanded to enable community pharmacists to prescribe adaptations (e.g., modify a dose or regimen) or prescribe a medication for a chronic disease including diabetes, asthma, and heart disease but not CKD unless associated with diabetes. Community pharmacists commonly see individuals with CKD. Interviews of Nova Scotia pharmacists recently revealed barriers to assessing kidney function, medication dosing and prescribing in CKD. These pharmacists emphasized the need to develop a collaborative, evidence and expert-informed drug dosing and decision support tool to optimize prescribing in the CKD population. Another study noted that prescribing by Nova Scotia community pharmacists significantly increased when a diagnosis was supported by a protocol . This finding was also identified in another survey of community pharmacists in Ontario. Nova Scotia is recognized as a national leader in enabling full scope of pharmacy practice. Community pharmacist prescribers are in an ideal position to support the safe use of medications needed to protect and preserve kidney function in individuals with CKD. While electronic tools for patients, hospital drug order entry technologies and a general ambulatory clinical pathway for managing CKD in another province have been developed to improve care of CKD patients, tools to optimize prescribing in patients with CKD are absent from the literature. Having a tool to support Nova Scotian community pharmacists could mitigate inappropriate drug exposure and harm or preserve kidney function through appropriate prescribing. This research will enable the pharmacist's full scope of practice as a prescriber in caring for individuals with CKD in Nova Scotia.

This research will use different ways to see how the digital dosing tool works at participating pharmacy locations, like checking how many people use it, how well it helps adjust doses, and asking patients for feedback. We'll follow a method called RE-AIM, which looks at how many people are reached, how well the tool works, how easy it is for people to use, how it's put into practice, and if it continues to be used over time.

ELIGIBILITY:
Inclusion Criteria:

* individuals with an eGFR < 60 mL/min/1.73m2 AND
* receiving at least 1 tool target medication

Exclusion Criteria:

* individuals on dialysis
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be individuals over the age of 18 years who have been diagnosed with chronic kidney disease (CKD). Specifically, participants will have an estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73m², which indicates the presence of CKD. These individuals will be receiving one of the 30 target medications prescribed via a digital dosing tool.
  Participants will be selected from a sample of patients attending 10-12 community pharmacy sites spread across the province. These pharmacies will act as the study's recruitment hubs, providing access to participants who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Intervention Success and Intervention Safety | After 6 months of tool introduction.
  Quantitative measures of the number and type of target medications changed by community pharmacists with the tool or not changed including reasons, the number of patients who accept or decline the medication change including reasons, the number of potential level of harm or clinical impact as described by the Cornish classification system, and the number of unexpected clinically significant adverse events from medication changes with the tool.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tran J, Shaffelburg C, Phelan E, Neville H, Lively A, Poyah P, Tennankore K, More K, Soroka S, Harpell D, Wilson JA. Community pharmacists' perspectives on assessing kidney function and medication dosing for patients with advanced chronic kidney disease: A qualitative study using the theoretical domains framework. Can Pharm J (Ott). 2023 Jul 7;156(5):272-281. doi: 10.1177/17151635231176530. eCollection 2023 Sep-Oct. PMID 38222892
- [Background] Wilson JA, Ratajczak N, Halliday K, Battistella M, Naylor H, Sheffield M, Marin JG, Pitman J, Kennie-Kaulbach N, Trenaman S, Gillis L. Medications for community pharmacists to dose adjust or avoid to enhance prescribing safety in individuals with advanced chronic kidney disease: a scoping review and modified Delphi. BMC Nephrol. 2024 Oct 29;25(1):386. doi: 10.1186/s12882-024-03829-y. PMID 39472832